CLINICAL TRIAL: NCT02825537
Title: Study of the Effect of Class III Elastic Venous Compression Focused on 33 mmHg on Water Balance Change in Healthy Subjects. Exploratory, Randomized, Open-label, Controlled and Crossover Study
Brief Title: Study of the Effect of Elastic Compression (French Class III) on Water Balance Change in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Innothera (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CVE101-15
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Stockings, Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With use of compression stocking (Experimental): Use of compression stocking during 3 consecutives days
  Interventions: Device: Compression stocking
- Without use of compression stocking (Other): No use of compression stocking during 3 consecutives days
  Interventions: Other: No use of compression stocking

INTERVENTIONS:
Device: Compression stocking — A class III (20 to 36 mm Hg) elastic compression stocking according to the french classification
  Arms: With use of compression stocking
Other: No use of compression stocking — No use of compression stocking
  Arms: Without use of compression stocking

SUMMARY:
The main objective of this study is to compare precisely, under standardized test conditions, water balance changes in healthy subjects with or without the daytime use of compression stocking.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject aged 40 years old or more,
2. Subject with a Body Mass Index (BMI) between 18.5 and 30 kg/m²,
3. Subject with a body fat percentage between 11 and 27 % of his weight, as measured by impedancemetry,
4. Subject with a muscle mass index of less than 55% of his weight, as measured by impedancemetry,
5. Subject with a water status, as measured by impedancemetry, between + / - 5 liters of his normal value, as indicated by the impedancemetry,
6. Healthy subject, registered in the French biomedical research volunteer national database,
7. Subject whose lower limb measurements correspond to the size grid of the compression stocking used,
8. Subject agreeing to abstain from alcohol intake during all hospitalization periods,
9. Subject practicing under 5 hours of intense physical activity per week, on average, in the 4 weeks preceding the screening visit (marathon training, military training ...),
10. Subject agreeing to abstain from any strenuous activity , especially sports, from the screening visit to the end of study (including during the out-patient period),
11. Subject accepting the constraints of the study,
12. Subject being available during the whole period of the study,
13. Subject who has signed the consent form after being adequately informed and receiving the information sheet,
14. Subject affiliated to the French social security system or receiving benefits of that type.

Exclusion criteria:

1. Subject who is a smoker or a former smoker who stopped smoking less than 6 months ago,
2. Subject following a salt-free diet,
3. Subject following or planning to follow a diet,
4. Subject having a temperature ≥ 38,5°C in the morning,
5. Subject having, upon clinical examination, a systolic blood pressure (SBP) < 91 mmHg or > 139 mmHg, a diastolic blood pressure (DBP) < 41 mmHg or > 89 mmHg, or a heart rate (HR) < 40 bpm or > 100 bpm, and judged clinically significant by the investigator,
6. Subject having an intestinal transit disorder that disrupts hydroelectric balance,
7. Alcohol-dependent subject or subject with a positive alcohol breath test,
8. Subject having a localized or general edema (a simple evening edema of the legs or ankles is accepted for inclusion),
9. Subject suffering from insulin-dependent or uncontrolled diabetes (controlled diabetes is accepted),
10. Subject with a serious, stabilized, or progressive illness (as judged by the investigator),
11. Subject with hypertension or heart failure,
12. Subject with known renal function disorders,
13. Subject with known liver failure,
14. Subject with venous insufficiency of clinical class C3, C4, C5 or C6 according to the Clinical / Etiological / Anatomical / Pathophysiological (CEAP) classification,
15. Subject following long-term therapy with diuretics, nonsteroidal anti-inflammatory drugs (NSAIDs), steroids, nutritional supplements or opiates,
16. Subject having, upon questioning or clinical examination, advanced peripheral neuropathy, skin infections, eczematous dermatitis, or weeping skin disorder of the leg,
17. Subject with a medical contraindication to compression therapy according to the interview or clinical examination: phlegmatia coerulea dolens, septic thrombosis, intolerance to the product including the self-supporting band, allergic reaction to any component, arteritis obliterans of lower limbs, advanced diabetic microangiopathy,
18. Subject with active implants, such as a pacemaker or other mechanical heart device , and non-active implants, for example a hip prosthesis (dental implants are authorized),
19. Subject who is participating in another clinical trial or who is in the exclusion period from a previous study,
20. Person deprived of freedom by judicial or administrative decision, or a person hospitalized without their consent,
21. Subject of legal age who is protected by law or under guardianship,
22. Subject with a current mental or psychiatric disorder or a history of mental or psychiatric disorder, or any other factor limiting the collection of informed consent,
23. Person who works for the Contract Research Organisation or for Innothéra laboratories, or has a dependent relationship with these entities.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evolution of the total bodily fluid volume in the daytime sequence measured by impedancemetry with or without daytime use of compression stocking | adjusted over 3 consecutive days

SECONDARY OUTCOMES:
Evolution of the water balance in daytime sequence,in night sequence and on a 24h sequence with or without daytime use of compression stocking | adjusted over 3 consecutive days
Evolution of the subject's weight (in kilograms), in daytime sequence, in night sequence and on a 24 h sequence with or without daytime use of compression stocking | adjusted over 3 consecutive days
Evolution of the volume of urine determined by weight (in kilograms),in daytime sequence, in night sequence and a 24h sequence with or without daytime use of compression stocking | adjusted over 3 consecutive days
Evolution days of the neck circumference (in centimeter) in a dynamic sequence, in supine sequence and on a 24h sequence with or without daytime use of compression stocking | adjusted over 3 consecutive days
Evolution of leg perimeters (in centimeter) in 3 points in dynamic sequence, in supine sequence , and over 24h sequence with or without daytime use of compression stocking | adjusted over 3 consecutive days
Evolution of the time and volume of the first urine after H0 determined by weight (in kilograms) with or without daytime use of compression stocking | adjusted over 3 consecutive days
Evolution of the quantity of NaCl excreted in urine in daytime sequence, in night sequence, and over 24 h sequence with or without daytime use of compression stocking | adjusted over 3 consecutive days
Evolution of the total bodily fluid volume in night sequence and on a 24h sequence measured by impedancemetry with or without daytime use of compression stocking | adjusted over 3 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Hakim Charfi, MD, Principal Investigator — Biotrial
Locations (1):
- Biotrial, Rennes, France